CLINICAL TRIAL: NCT00950378
Title: Non-Invasive Management of Chronic Venous Insufficiency
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: PhiloMetron, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 27610; 1R43HL092673 (NIH); University of Utah (Other Grant/Funding Number: 54901268)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Venous Insufficiency
Keywords: edema; blood supply; lower legs; venous stasis
MeSH Terms: conditions — Venous Insufficiency; Edema; Varicose Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CVI: Varicose veins, varicose veins with leg swelling, venous stasis skin color changes, no open ulcers
- No treatment: Subjects with no venous disease CEAP (clinical etiology antomy pathophysiology)Class 0

SUMMARY:
The purpose of this study is:

-item one to use two new non-invasive technologies to evaluate scarring and swelling associated with chronic venous insufficiency.

The study hypothesis:

- item one non-invasive technologies can provide a tool for assessing risk of ulcer development based on the tissue edema and alteration.

ELIGIBILITY:
Inclusion Criteria:

* participants with CVI with CEAP class 4 or higher
* participants with no CVI class 0

Exclusion Criteria:

* open ulcers or lower extremity amputation
* diabetics with HbA1C greater than 7.0
* arterial occlusive disease
* BMI greater than 35
* any connective tissue disorder (lipodermatosclerosis and fibrosis)
* participants with metallic prosthesis or implants
* participants with renal impairment
* pregnancy
* inability or refusal to wear compression stockings prescribed by physician (CVI patients only)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: CVI subjects will be recruited from University of Utah vascular surgery service.Control group will be recruited from the community.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-07; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To provide device development to assess tissue changes associated with chronic venous insufficiency | two years

SECONDARY OUTCOMES:
To compare device development to existing clinical measurement | two years

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Hopf, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Eberhardt RT, Raffetto JD. Chronic venous insufficiency. Circulation. 2005 May 10;111(18):2398-409. doi: 10.1161/01.CIR.0000164199.72440.08. No abstract available. PMID 15883226
- [Background] Olin JW, Beusterien KM, Childs MB, Seavey C, McHugh L, Griffiths RI. Medical costs of treating venous stasis ulcers: evidence from a retrospective cohort study. Vasc Med. 1999;4(1):1-7. doi: 10.1177/1358836X9900400101. PMID 10355863